CLINICAL TRIAL: NCT00002120
Title: Randomized Phase I Study of Trimetrexate Glucuronate (TMTX) With Leucovorin (LCV) Protection Plus Dapsone Versus Trimethoprim / Sulfamethoxazole (TMP/SMX) for Treatment of Moderately Severe Episodes of Pneumocystis Carinii Pneumonia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Bioscience (Industry)
Collaborators: Jacobus Pharmaceutical (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 224A; TMTX A009
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; Trimetrexate; Pneumonia, Pneumocystis carinii; Leucovorin; Dapsone; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — trimetrexate glucuronate; Trimethoprim; Sulfamethoxazole; Dapsone; Leucovorin

INTERVENTIONS:
Drug: Trimetrexate glucuronate
Drug: Trimethoprim
Drug: Sulfamethoxazole
Drug: Dapsone
Drug: Leucovorin calcium

SUMMARY:
To evaluate the safety of the combination of trimetrexate glucuronate (TMTX) and dapsone with leucovorin protection versus trimethoprim/sulfamethoxazole (TMP/SMX) in patients with AIDS and moderately severe Pneumocystis carinii pneumonia (PCP). To determine the pharmacokinetic parameters of TMTX, leucovorin, and dapsone and of TMP/SMX when given to patients with AIDS and moderately severe PCP.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Empiric therapy for other opportunistic pulmonary infection (TB or fungi) for the first 72 hours of study enrollment ONLY, until presence of suspected pathogens can be confidently excluded.

Patients must have:

* AIDS.
* Confirmed diagnosis of PCP.
* Alveolar-arterial differences in dissolved oxygen >= 35 mm Hg but < 55 mm Hg on room air.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Severe renal or hepatic dysfunction.
* Serious or life-threatening intolerance to TMP/SMX, TMTX, or dapsone.
* Concurrent pneumothorax.
* Active pulmonary tuberculosis or other inadequately treated opportunistic pulmonary infection (e.g., Cryptococcus neoforms, CMV). NOTE:
* Identification of Mycobacterium avium or CMV in sputum or BAL fluid does not exclude, since these organisms may be present without causing disease.
* Pulmonary Kaposi's sarcoma.
* Active opportunistic infections or malignancies requiring induction therapy with bone marrow suppressive drugs (e.g., ganciclovir) or hepatotoxic drugs (e.g., chemotherapy).
* Unable to have arterial blood gases on room air obtained at baseline.
* Unwilling to undergo bronchoscopy, if sputum induction does not reveal Pneumocystis carinii.
* Suspected malabsorption (e.g., ileus or severe diarrhea with > 6 stools/day).
* Known absence of G6PD activity.
* Large volume (1.0 to 1.5 liters) of intravenous fluid (5 percent in water) per 24 hours is medically inadvisable.
* Unwilling to comply with study design.

Concurrent Medication:

Excluded:

* Induction therapy with bone marrow suppressive drugs (e.g., ganciclovir) or hepatotoxic drugs (e.g., chemotherapy).
* AZT, ddI, ddC, d4T, or other antiretroviral therapy.

Patients with the following prior condition are excluded:

Prior history of serious or life-threatening intolerance to TMP/SMX. (NOTE:

* Patients with less severe reactions may be included at the discretion of the investigator and primary care provider.)

Prior Medication:

Excluded:

* More than 24 hours of systemic anti-PCP therapy within 2 weeks prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles County / Health Research Assoc / Drew Med Ctr, Los Angeles, California, United States